CLINICAL TRIAL: NCT05202444
Title: Evaluation of Using Piezoelectric Device Versus Conventional Saw for Osteotomy in Maxillary Orthognathic Surgery
Brief Title: The Use of Piezoelectric Surgery for Osteotomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Collaborators: Dar Al Shifa Hospital (Other)
Responsible Party: Principal Investigator, Abdullah Hammuda, Associate Professor, Suez University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 281
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Maxillofacial, Osteotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteotomy using piezoelectrical device (Experimental)
  Interventions: Procedure: Osteotomy using piezoelectrical device
- Osteotomy using surgical saw (Active Comparator)
  Interventions: Procedure: Osteotomy using piezoelectrical device

INTERVENTIONS:
Procedure: Osteotomy using piezoelectrical device — osteotomy were utilized using piezoelectric from device (Woodpeker) with its internal irrigation system. We used US2 tip using the maximum bone cutting program and maximum irrigation program for lateral maxillary wall osteotomy and USIR tip for the posterior maxillary wall osteotomy.
  The pterygoid osteotome was placed between the tuberosity and pterygoid plates while the hamulus is palpated palatally with the index finger to guide the osteotome direction preventing palatal perforation.With the pterygoid osteotome still in position, we used a thin osteotome to complete the osteotomy of the posterior wall of the maxilla.

SUMMARY:
Piezo-surgery was ﬁrst used in oral and maxillofacial surgery in 2001 by Vercellotti and colleagues to simplify maxillary sinus surgery by avoiding perforation of the schneiderian membrane. Later on ultrasonic bone cutting has been used in orthognathic procedures, extraction of impacted third molars , cyst enucleation, implant site preparation, temporomandibular join surgery , corticotomy-facilitated orthodontics, and head and neck oncological and reconstructive surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged from 18 to 35 years.
2. Patients were not suffering from systemic diseases that compromise wound or bone healing.
3. Patients indicated for leforte I or maxillary subapical osteotomy.
4. Patients agree the informed consent .

Exclusion Criteria:

1. Patients suffering from systemic disease that may affect bleeding or bone healing
2. Syndromicdentofacial deformity patients.
3. Patients were subjected to previous maxillary orthognathic surgery.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Intra-operative Bleeding | From begining of the surgery till the end
Osteotomy Time | From begining of the surgery till the end

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided